CLINICAL TRIAL: NCT05354635
Title: Therapeutic Follow-up of Antibiotics in Pediatric Intensive Care
Acronym: STAR-P
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/CHU/05
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Intensive Care Units, Pediatric

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Antibiotics Dosing — Dosing concerns the main antibiotics used in the unit: b-lactams, linezolid, vancomycin and aminosides

SUMMARY:
Currently, recommendations for antibiotic testing (ATS) in adult intensive care have been published. The 2018 SFAR and the Abdul- Aziz et al expert conference recommend routine testing for β-lactams, aminoglycosides, linezolid, and vancomycin and provide plasma concentration goals. No recommendations have been made for the pediatric intensive care unit (PICU) population. However, several articles report suboptimal plasma concentrations for the most frequently used antibiotics in PICU. The University Hospital of Reunion is the reference center for the western region of the Indian Ocean. This region presents a large mixed population due to the migratory flow, as well as a specific bacterial ecology. This suggests that the data already collected on antibiotic dosage in other European studies may not be fully extrapolated to Reunion Island.

It is in this context that we will study the plasma concentration of antibiotics for all children who received the most commonly used antibiotics (β-lactams, linezolid, vancomycin, and aminoglycosides) during their hospitalization in PICU.

ELIGIBILITY:
Inclusion Criteria:

* Any child hospitalized in the pediatric intensive care unit of the CHU Nord de La Réunion,
* Age is less than 18 years,
* Having started a curative antibiotic therapy by β-lactam, linezolid, vancomycin or aminosides.
* For whom a non-opposition has been collected orally from both or one of the child's legal guardians and from the child himself (if applicable),
* Covered by Social Security.

Exclusion Criteria:

-Patients on prophylactic antibiotic therapy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The aim of the research is to evaluate the adequacy of antibiotic therapy in children admitted to the pediatric intensive care unit at the University Hospital of La Réunion. The study population is intended to be exhaustive and will include all subjects affiliated to the Social Security who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The occurrence of at least one "underdosing" event of one of the Antibiotics used in a patient included during his or her hospitalization in pediatrics intensive care unit (PICU) | 2 months
  Underdosing is defined as a measurement of plasma concentration below the optimal therapeutic concentration (OTC)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Denis, Reunion

IPD SHARING:
Plan to Share IPD: No